CLINICAL TRIAL: NCT03722667
Title: The Effects of Technology-based Intervention and Positive Psychological Training on Cognitive Processing and Blood Pressure Control in African Americans
Brief Title: Technology-based Intervention and Positive Psychological Training for Blood Pressure Control in African Americans
Acronym: TechSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Still, Assistant Professor, Frances Payne Bolton School of Nursing, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5P30NR015326-05 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Self-management; Technology
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The investigators hypothesize that African Americans' hypertension self-management behaviors are influenced by the ability of the individual to task differentiate between the DMN and TPN neural processing. Furthermore, such behaviors will lead to improved BP control and HRQoL. Using a two-arm RCT pilot study, investigators will compare the effects of TechSuPPorT and the Technology-based component arm on BP, HRQoL, and psychological health (affective well-being, depressive symptoms, anxiety) and cognitive task differentiation of the DMN and TPN neural networks. Data will be collected at three points: baseline, 8 weeks and 12 weeks. Brain scans (fMRIs) will be captured at baseline and following the intervention at 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Based Component (Placebo Comparator): A Technology-based interventions comprised of three technolgy components accessible via smartphone to support self-managing hypertension.
  Interventions: Behavioral: Technology-based Component
- TechSupport (Experimental): A Technology-based interventions comprised of three technolgy components plus positive psychological training accessible by smartphone to support self-managing hypertension.
  Interventions: Behavioral: TechSupport

INTERVENTIONS:
Behavioral: Technology-based Component — This intervention is comprised of three technology components: a) six weekly web-based modules focused on improving knowledge and skills to manage hypertension; (b) personalized medication adherence support (SMS reminder messages, adherence feedback, health and lifestyle tips) through Medisafe app; and (c) self-monitoring blood pressure to support self-managing hypertension.
  Arms: Technology-Based Component
Behavioral: TechSupport — The TechSupport intervention is the combination of both an behavioral and emotional intervention.
  Technology-based Components: This intervention is comprised of three technology components: a) six weekly web-based modules focused on improving knowledge and skills to manage hypertension; (b) personalized medication adherence support (SMS reminder messages, adherence feedback, health and lifestyle tips) through Medisafe app; and (c) self-monitoring blood pressure to support self-managing hypertension.
  Positive Psychological Training (PPT): This intervention will include a structured online training and skill building for PPT accessible by smartphone on techniques to promote optimism, resilience, well-being, and self-confidence.
  Arms: TechSupport

SUMMARY:
The purpose of this pilot study is to evaluate the effects of a theoretically-derived technology-based intervention (called TechSuPPorT) and its associated neurological mechanisms for hypertension self-management in African Americans.

The investigators will compare two intervention arms in this study, the Technology-Based Component Only arm (comparison group) and the TechSuPPorT arm (intervention group) in 20 African Americans with uncontrolled hypertension. We aim to:

1. Determine whether there are differences in blood pressure (BP), health-related quality of life (HRQoL), and psychological health (affective well-being, depressive cognitions, anxiety) betweenTechSuPPorT and the Technology-based Component only arm.
2. Determine whether there are differences in self-management behaviors (medication adherence, diet, exercise, self-monitoring BP) between the two groups.
3. Examine whether self-efficacy, decision-making, motivation, patient activation, and perceived stress, and positive emotions mediate the relationship between the interventions and self-management behaviors.
4. Determine if social support, demographics (age, gender, education), discrimination, and technology utilization moderate self-management behaviors, BP, HRQoL, and psychological health.
5. Explore differences in neural processing (diffusion tensor imaging [DTI]/ task positive network [TPN] task-differentiation), and stress response (cortisol and inflammation panel) between the two groups.

DETAILED DESCRIPTION:
The investigators will conduct a two-arm randomized clinical trial to compare the effects of an Technology-Based Component Only arm and TechSuPPorT on self-management behaviors, BP control, and HRQoL outcomeson cognitive task switching between the DMN and TPN neural networks using Functional Magnetic Resonance Imaging (fMRI) and Diffusion Tensor Imaging (DTI). Both groups will be exposed to the three Technology-based components: (a) six weekly web-based modules focused on improving African Americans' knowledge and skills of hypertension management; (b) personalized medication adherence support (SMS reminder messages, adherence feedback, health and lifestyle tips) through Medisafe, a smartphone app; and (c) self-monitor BP with study provided BP monitor. Participants in the TechSuPPorT arm will receive the three Technology-based components plus positive psychological training, a structured online training and skill building techniques to promote optimism, resilience, well-being, and self-confidence.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* 25 years and older
* diagnosed with hypertension defined, as BP ≥ 130/80 mmHg
* Taking at least one antihypertensive medication(s)
* own an android smartphone
* able to read and understand English

Exclusion Criteria:

* are unable to give informed consent or judged to have impaired cognitive ability or severe memory deficits
* currently practicing positive psychological training
* have a history of medical conditions or procedures that is contraindicated for fMRI scanning (cardiac pacemaker, sternal wires, or metal implants)
* have a history of claustrophobia requiring anxiolytics or sedation
* pregnant at time of enrollment

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Baseline to 8 weeks and 12 weeks
  Measure of participants' in clinic blood pressure (average of three blood pressure readings)
PROMIS Global Health-10 [health-related quality of life] | Baseline to 8 weeks and 12 weeks
  Change in total summed score on PROMIS Global Health-10. Higher scores indicate greater health-related quality of life. Range is 4-20.
PROMIS Short Form, Positive Affect -15a [positive affect and well-being] | Baseline to 8 weeks and 12 weeks
  Change in total summed score on PROMIS Short Form, Positive Affect 15a. Higher scores indicate greater positive affect and well being. Range is 15-45.
PROMIS- 29, Depression Subscale 4a [depressive symptoms] | Baseline to 8 weeks and 12 weeks
  Change in total summed PROMIS-29, Depression Subscale 4a. Higher scores indicate greater depressive symptoms. Range is 4 to 20.
PROMIS- 29, Anxiety Subscale 4a [anxiety symptoms] | Baseline to 8 weeks and 12 weeks
  Change in total summed PROMIS-29, Anxiety subscale. Higher scores indicate greater anxiety. Range is 4-20.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn H Still, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Still CH, Jack AI, Wright KD, Sattar A, Moore SM. Neural Processing of Health Information and Hypertension Self-Management in African Americans. Nurs Res. 2022 Jul-Aug 01;71(4):303-312. doi: 10.1097/NNR.0000000000000592. Epub 2022 Mar 18. PMID 35302958
- [Derived] Still CH, Margevicius S, Harwell C, Huang MC, Martin L, Dang PB, Wright Jnr JT. A Community and Technology-Based Approach for Hypertension Self-Management (COACHMAN) to Improve Blood Pressure Control in African Americans: Results from a Pilot Study. Patient Prefer Adherence. 2020 Nov 23;14:2301-2313. doi: 10.2147/PPA.S283086. eCollection 2020. PMID 33262580